CLINICAL TRIAL: NCT02010476
Title: Cerebrospinal Fluid Changes in Insulin-Resistant Men
Brief Title: Alzheimer's Disease Biomarkers in Cerebrospinal Fluid in Insulin-resistant Men
Acronym: ADDM
Status: Completed | Type: Observational
Sponsor: University of Eastern Finland (Other)
Collaborators: King's College London (Other); Sahlgrenska University Hospital (Other); Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Hilkka Soininen, Professor, University of Eastern Finland
Other Study IDs: 3971
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease, CSF biomarkers, Insulin resistance
MeSH Terms: conditions — Alzheimer Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, white cells, urine, cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal insulin sensitivity: cognitively normal men without insulin resistance
- Insulin resistance: cognitively normal men with insulin resistance

SUMMARY:
Type 2 diabetes mellitus has been associated with an about 2-fold increase in risk of Alzheimer's disease (AD). Patients with AD have been reported to have reduced insulin sensitivity. It may be hypothesized that, compared to insulin sensitive subjects otherwise similar in general health and body habitus, insulin resistant subjects are more likely to have cerebrospinal fluid (CSF) indicators of incipient AD pathology, abnormalities in CSF peptides related to insulin signaling and glucose homeostasis, and possibly other metabolites that are associated with a risk of AD. The objective of this study is to examine the relation of insulin resistance and the concentrations of CSF biomarkers. The results of this study may be useful in the detection of the subjects who are at risk for cognitive decline and AD.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus has been associated with an approximately 2-fold increase in risk of Alzheimer's disease (AD). Patients with AD have been reported to have reduced insulin sensitivity, and to have insulin concentrations that are elevated in plasma and decreased in cerebrospinal fluid (CSF). Cognitively normal individuals with insulin resistance are thus of interest in our effort to gain an understanding of the antecedents of this problem. It may be hypothesized that, compared to insulin sensitive subjects otherwise similar in general health and body habitus, insulin resistant subjects are more likely to have CSF indicators of incipient Alzheimer pathology, abnormalities in CSF peptides related to insulin signaling and glucose homeostasis, and possibly other metabolites that are associated with a risk of AD.

The objectives are to 1) assess the concentrations of biomarkers of Alzheimer pathology in the CSF of cognitively normal men with and without insulin resistance, and 2) assess the concentrations of other CSF biomarkers of potential relevance to insulin resistance and AD in the CSF of cognitively normal men with and without insulin resistance.

All subjects with eligibility will have had an oral glucose tolerance test performed within the past 3 months that revealed a normal fasting blood level and normal glucose tolerance. In addition, they will have had no history of significant cognitive disorders, no prior diagnosis of diabetes mellitus, and will not be receiving insulin or oral hypoglycemic. Eligibility for inclusion in the insulin-resistant group will be defined by scores on the Matsuda Index; non-insulin resistant controls will have normal values on the Matsuda Index. An effort will be made to ensure that both groups (i.e., those with insulin resistance and those without insulin resistance) will be similar in age, weight, BMI, and Apo E4 genotype (APOE).

All procedures will be performed on a single visit. The subjects will undergo a Mini-Mental Status Examination (MMSE) performed by a qualified examiner. In addition, a blood sample will be obtained for measurements of basic blood chemistry (electrolytes, creatinine, glucose, total protein, and albumin), hematology, thyroid function, metabolic function (e.g. fasting plasma glucose and insulin levels) and for proteomic analysis. The APOE genotype will be determined from the blood samples, if it has not been assessed earlier. A lumbar puncture will be performed to obtain CSF samples that will be used to determine concentrations of biomarkers of AD pathology and to find out new biomarkers that may reflect AD pathology.

All materials will be used according to national ethical guidelines for Good Clinical Practice. Analyses of the CSF for levels of beta-Amyloid biomarkers, total tau and phosphorylated tau will be done using a sandwich ELISA. Descriptive statistics will be provided for each analyte, comparing the 2 groups of subjects.

All participants will provide written informed consent. Blood and CSF samples will be analysed also by collaborators in other European countries. Before analysis and sending data and blood/CSF samples to partners of the project, all clinical information and sample information will be made anonymous (coded data). Personal information, i.e., name and personal identity number, is removed from data/samples, and separate codes are given to them before delivering them to other partners for the purposes of the project. Methods for database maintenance and data delivery will be used that have proved to be functional in previous research projects. A formal description of the different data formats, access routines and tools for basic processing will be created at the start of the project.

ELIGIBILITY:
Inclusion Criteria:

* Males 55-70 years in age
* Normal cognitive function, as evidenced by the following: 1. Living independently in the community, 2. No memory complaints; Score on Mini Mental State Examination >= 25 (Folstein 1975), 3. Score on Functional Activities Questionnaire < 9
* Has had oral glucose tolerance test including determination of plasma glucose and insulin levels at baseline and 30 and 120 minutes within the past 3 months, meeting the following criteria: 1. Normal fasting blood glucose (<7.0 mmol/l), 2. Normal glucose tolerance at 120 minutes (<11.1 mmol/l), 3. Meets criteria for either normal insulin sensitivity or insulin resistance, based upon the Matsuda insulin sensitivity index
* Willing to have lumbar puncture

Exclusion Criteria:

* Evidence of significant neurological disease, including 1. Abnormal neurological examination, 2. History of stroke (other than lacunar infarction), 3. prior diagnosis of mild cognitive impairment, significant head injury with impairment of consciousness > 24h, brain tumor, multiple sclerosis, epilepsy, or hydrocephalus, 4. Diagnosis or family history consistent with autosomal dominantly inherited AD
* Prior diagnosis of diabetes mellitus type 1 or 2
* Evidence of significant metabolic or endocrine disorder associated with risk of cognitive impairment, e.g., hypothyroidism or B12 deficiency
* Major psychiatric disorder, including psychosis
* Evidence of significant systemic disease, including: congestive heart failure, renal failure, hepatic cirrhosis, significant chronic obstructive pulmonary disease, cancer within the past 5 years (other than nonmetastatic basal cell and squamous cell carcinoma of the skin)
* Excluded concomitant medications: 1. Acetylcholinesterase inhibitors, Memantine (Alzheimer's disease medications), 2. Insulin or oral hypoglycemics, 3. Anticoagulants (excluding aspirin, clopidogrel, dipyridamole, or other antiplatelet drugs), 4. Neuroleptic drugs, including risperidone, olanzapine, quetiapine, and ziprasidone, 5. Receipt of an investigational drug within the past 30 days (or within 5 half-lives of an investigational drug, whatever is longest)

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the research data sources of METSIM study (METabolic Syndrome In Men; professor Markku Laakso) performed in the Department of Internal Medicine, University of Eastern Finland
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Abnormal concentrations of CSF biomarkers related to Alzheimer's disease | during a single visit, i.e., day 1

SECONDARY OUTCOMES:
Abnormal concentrations of other CSF biomarkers of potential relevance to insulin resistance and Alzheimer's disease | during a single visit, i.e., day 1

CONTACTS AND LOCATIONS:
Overall Officials: Hilkka Soininen, Professor, Principal Investigator — University of Eastern Finland
Locations (1):
- Department of Neurology and Brain Research Unit, Institute of Clinical Medicine, University of Eastern Finland, Kuopio, Finland